CLINICAL TRIAL: NCT07045987
Title: FUtile Reperfusion in acuTe iscHEmic stRoke- FURTHER
Brief Title: Exploration and Establishment of an Early Warning System for Futile Reperfusion - A I S
Status: Enrolling by invitation | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: National Science and Technology Major Project (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY20252127
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke (AIS); Endovascular Thrombectomy; Neurovascular Unit- Brain Lymphatic System
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort registration study is to establish an early warning system for futile recanalization in acute ischemic stroke by analyzing multi-omics information to identify key regulatory nodes and target molecules in ineffective recanalization.

The core issue addressed by this research is: Identifying key regulatory nodes and target molecules closely associated with futile recanalization, revealing the interactions among the neurovascular unit, peripheral immune cells, and the brain lymphatic system, as well as developing early diagnostic biomarkers and novel diagnostic technologies for futile recanalization.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged ≥18 years 2. Acute ischemic stroke confirmed by clinical and neuroimaging criteria (CT or MRI) 3. Clinical indication for thrombectomy 4. Provision of signed informed consent

Exclusion Criteria:

* 1. Preexisting dementia or severe disability (modified Rankin Scale score ≥3) 2. Cerebral vascular malformations, neoplasms, abscesses, or other significant non-ischemic brain pathologies 3. Life-limiting systemic comorbidities (e.g., end-stage organ failure, metastatic malignancies) with anticipated survival <6 months 4. Patient or legally authorized representative declined consent 5. Anticipated poor protocol adherence or loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18y) with thrombectomy-eligible acute ischemic stroke confirmed by neuroimaging, meeting prespecified inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
3-month mRS score | From enrollment to the end of treatment at 3 months

OTHER OUTCOMES:
All-cause mortality within 3 months | From enrollment to the end of treatment at 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Luojun WANG, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hussein HM, Georgiadis AL, Vazquez G, Miley JT, Memon MZ, Mohammad YM, Christoforidis GA, Tariq N, Qureshi AI. Occurrence and predictors of futile recanalization following endovascular treatment among patients with acute ischemic stroke: a multicenter study. AJNR Am J Neuroradiol. 2010 Mar;31(3):454-8. doi: 10.3174/ajnr.A2006. Epub 2010 Jan 14. PMID 20075087
- [Background] Liu X, Dai Q, Ye R, Zi W, Liu Y, Wang H, Zhu W, Ma M, Yin Q, Li M, Fan X, Sun W, Han Y, Lv Q, Liu R, Yang D, Shi Z, Zheng D, Deng X, Wan Y, Wang Z, Geng Y, Chen X, Zhou Z, Liao G, Jin P, Liu Y, Liu X, Zhang M, Zhou F, Shi H, Zhang Y, Guo F, Yin C, Niu G, Zhang M, Cai X, Zhu Q, Chen Z, Liang Y, Li B, Lin M, Wang W, Xu H, Fu X, Liu W, Tian X, Gong Z, Shi H, Wang C, Lv P, Tao Z, Zhu L, Yang S, Hu W, Jiang P, Liebeskind DS, Pereira VM, Leung T, Yan B, Davis S, Xu G, Nogueira RG; BEST Trial Investigators. Endovascular treatment versus standard medical treatment for vertebrobasilar artery occlusion (BEST): an open-label, randomised controlled trial. Lancet Neurol. 2020 Feb;19(2):115-122. doi: 10.1016/S1474-4422(19)30395-3. Epub 2019 Dec 9. PMID 31831388
- [Background] Ma H, Che R, Zhang Q, Yu W, Wu L, Zhao W, Li M, Wu D, Wu C, Ji X. The optimum anticoagulation time after endovascular thrombectomy for atrial fibrillation-related large vessel occlusion stroke: a real-world study. J Neurol. 2023 Apr;270(4):2084-2095. doi: 10.1007/s00415-022-11515-y. Epub 2023 Jan 3. PMID 36596867
- [Background] Dong Q, Dong Y, Liu L, Xu A, Zhang Y, Zheng H, Wang Y. The Chinese Stroke Association scientific statement: intravenous thrombolysis in acute ischaemic stroke. Stroke Vasc Neurol. 2017 Jun 2;2(3):147-159. doi: 10.1136/svn-2017-000074. eCollection 2017 Sep. PMID 28989804
- See also: Related Info — https://doi.org/10.1007/s00234-018-2016-2
- See also: Related Info — https://doi.org/10.1186/s42466-022-00215-7
- See also: Related Info — https://doi.org/10.1136/neurintsurg-2020-015889